CLINICAL TRIAL: NCT06291974
Title: Efficacy of Solid Versus Ground Reaction Ankle Foot Orthosis on Muscular Activity in Children With Spastic Diplegic in Cerebral Palsy
Brief Title: Ankle Foot Orthosis on Muscle Activity in Cerebral Palsy
Status: Not yet recruiting | Type: Observational
Sponsor: Delta University for Science and Technology (Other)
Responsible Party: Sponsor
Other Study IDs: delta2024
Record Dates: First submitted 2024-02-20; First posted 2024-03-04 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-02

CONDITIONS: Cerebral Palsy Spastic Diplegia
MeSH Terms: conditions — Cerebral Palsy | interventions — Electromyography

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

INTERVENTIONS:
Diagnostic Test: electromyography — Surface Electromyography (SEMG) is a measurement of the electrical activity in muscles as a byproduct of contraction.
  It is the summation of action potentials from the muscle fibers under the electrodes placed on the skin

SUMMARY:
To compare the effect of solid ankle foot orthosis and ground reaction foot orthosis on the muscle activity in children with spastic diplegic cerebral palsy (Gross Motor Functional Classification Scale III).

DETAILED DESCRIPTION:
Few studies have examined muscular activity via electromyography (EMG) during quiet standing in children with cp.

A few studies have examined the benefits of ground reaction ankle foot orthosis, showing that it could effectively reduce or eliminate the crouch position in children with spastic cerebral palsy however little is known about the benefits of GRAFOs on postural control mechanisms in static standing in children with CP.

Previous Studies suggested that appropriate tuning of ankle foot orthosis properties may reduce muscle demand for children with CP.

So, this study may be a guide in management of postural instability in children with spastic diplegic cerebral palsy in standing position.

ELIGIBILITY:
Inclusion Criteria:

* Spasticity level II in lower limb muscles according to Modified Ashworth Scale.
* Able to follow order.
* Aged from 6 to 12 years old.

Exclusion Criteria:

* Visual or obvious detected vestibular sensory disorders or cerebellar disease.
* Botox injection in the last 6 months.
* Cognitive deficits or disturbed conscious level.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: children diagnosed with cp spastic diplegia with postural instability will represent the sample of this study.
  They will be selected from the clinic of faculty of physical therapy, delta university and my private clinic.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-03-15 (Estimated); Primary Completion 2024-10-15 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
muscle activity by Electromyography device | up to 12 months
  activity of gastrocnemius ad tibialis anterior muscle by Electromyography device